CLINICAL TRIAL: NCT03942965
Title: Multi-center Prospective Registry Study Utilizing a Double Balloon Accessory Device to Facilitate Endoscopic Polypectomy in Large Intestine.
Brief Title: Registry Evaluation of a Double Balloon Accessory Device
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lumendi, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DD_20
Record Dates: First submitted 2019-05-03; First posted 2019-05-08 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Adenomatous Polyp of Colon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Double balloon accessory device — Double balloon accessory device is used during the endoscopic polypectomy procedure
  Other Names: DiLumen

SUMMARY:
This study is collecting standard of care information pertaining to the use of the accessory device and patient outcomes when this double balloon accessory device is used during endoscopic procedures in the colon.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for endoscopic removal of suspected adenomatous benign polyps(s)
2. Patients capable of giving informed consent in English
3. No medical contraindication to endoscopic mucosal resection or endoscopic submucosal disection

Exclusion Criteria:

1. No patients less than 18 years of age.
2. Any contraindication to colonoscopy with due to subject's colon anatomy (i.e. stricture)
3. History of open or laparoscopic colorectal surgery
4. History of Inflammatory Bowel Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigator's practice
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Ability to perform the procedure safely and effectively with the study device. | Intraoperatively
  Investigator answers yes or no

SECONDARY OUTCOMES:
Time to reach target lesion | Intraoperatively
  Time measurement in hours and minutes
Time to remove lesion after intervention begins | Intraoperatively
  Time measurement in hours and minutes
Total time using study device during case | Intraoperatively
  Time measurement in hours and minutes
Total case time | Intraoperatively
  Time measurement in hours and minutes
Total defect closure time | Intraoperatively
  Time measurement in hours and minutes
User feedback on device performance | Intraoperatively
  Investigator rates the ease of use (easy, somewhat easy, somewhat difficult and difficult) of the device.
Number of Study Subjects with Treatment Related Adverse Events | Up to 30 days
  No moderate to severe mucosal injury, perforations or bleeding related to the use of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida - Division of Gastroenterology, Hepatology and Nutrition, Gainesville, Florida
  - Geisinger Health System, Danville, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No